CLINICAL TRIAL: NCT02301884
Title: Open-labeled Pilot Study of Intralymphatic Immunotherapy (ILIT) for House Dust Mite, Cat, and Dog Allergen in Allergic Rhinitis Patients
Brief Title: Pilot Study of Intralymphatic Immunotherapy (ILIT) for House Dust Mite, Cat, and Dog Allergen in Allergic Rhinitis
Acronym: pILIT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Principal Investigator, Sang Min Lee, Assistant professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBIRB2013-35
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Allergens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allergen extract (Experimental): Causal allergen such as D. farinae (30 AU/ml), D. pteronyssinus (30 AU/ml), cat hair (10 AU/ml), dog hair/dander (1:1/10 w/v), or combination of those.
  Allergen extract, HollisterStier, New Orleans, USA. Intralymphatic injection in volume of 0.1 ml, three times with 4-week interval. Concentration was increased, decreased, or unchanged at 2nd or 3rd injection according to local or systemic reaction after previous injection
  Interventions: Biological: Allergen extract

INTERVENTIONS:
Biological: Allergen extract — Causal allergen extract such as D. farinae, D. pteronyssinus, cat hair, dog hair/dander, or combination of those

SUMMARY:
The investigators performed open-labeled pilot study which evaluates the efficacy and safety of allergen-specific intralymphatic immunotherapy (ILIT) for allergens including Dermatophagoides farinae (Df), Dermatophagoides pteronyssinus (Dp), cat, and dog that are sensitized and provoke rhinitis-related symptoms in patients with allergic rhinitis.

DETAILED DESCRIPTION:
After informed consent, causal allergen was injected into inguinal lymph node through guidance by ultrasonography three times with 4-week interval. Initial dose of allergen was 1,000-fold diluted solution from maximal concentration of allergen extract for subcutaneous immunotherapy (30 AU/ml for Df or Dp, 10 AU/ml for Cat hair, and 1:1/10 weight/volume for dog hair/dander, HollisterStier, New Orleans, USA) in volume of 0.1ml. After the first dose, allergen concentration was escalated 3-fold at second dose, and 10-fold at third dose if there was no or mild local or systemic hypersensitivity reaction. The allergen concentration did not change at second or third dose if there was moderate local or systemic reaction. The allergen concentration was decreased by 10 or 100-fold from previous concentration if there was severe local or systemic reaction.

The investigators evaluated parameters regarding allergic rhinitis within a week before the first injection and 4 months after the first injection. These parameters included Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) and Sino-Nasal Outcome Test (SNOT-20), and Visual analogue scale (VAS) of symptoms including rhinorrhea, sneezing, nasal obstruction, postnasal drip, eye/nose/ear/palate itching, dyspnea, wheezing, chest discomfort as well as urticaria, angioedema, and itching on exposed skin during exposure to causal allergen in daily life. Skin prick test, intradermal test, blood sampling for serum allergen-specific IgE, exhaled nitric oxide, and nasal lavage for Th1, Th2, and Treg cytokines were also included. Adverse events were recorded and graded according to Muller's classification and Ring and Messmer's classification.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis to house dust mite (Df, Dp), cat or dog
* More than 3mm reaction at skin prick test for Df, Dp, cat or dog or more than class 3 at serum specific IgE level (UNICAP or MAST)

Exclusion Criteria:

* Uncontrolled or severe asthma according to Global Initiative of Asthma (GINA) guideline
* FEV1 less than 50% of predicted value if there is comorbid asthma
* Subject rejects the enrollment into study
* Low compliance
* Pregnancy or lactation
* Significant cardiovascular, hepatic, renal, hematologic, oncologic, or infectious diseases
* Administration of beta blocker, angiotensin converting enzyme inhibitor, tricyclic antidepressant, immunosuppressant including systemic glucocorticosteroid (20mg or more dose of prednisolone or equivalent dose of other steroid) within last 2 weeks
* Prior history of allergen-specific immunotherapy
* Allergic rhinitis caused by other perennial or seasonal allergen
* Vulnerable volunteer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
RQLQ | Baseline and 4 months after the first injection
  Rhinoconjunctivitis Quality of Life Questionnaire

SECONDARY OUTCOMES:
SNOT-20 | Baseline and 4 months after the first injection
  Sino-Nasal Outcome Test-20
Skin reactivity | Baseline and 4 months after the first injection
  Allergen/histamine ratio of mean wheal diameter in skin prick test, and allergen/saline ratio of mean wheal diameter in intradermal test
Serum total and allergen-specific IgE and IgG4 level | Baseline and 4 months after the first injection
  Serum total and allergen-specific IgE and IgG4 level using UNICAP, Thermofisher Scientific, Sweden
Nasal reactivity | Baseline and 4 months after the first injection
  Symptom score and volume 2-6 cm in acoustic rhinometry during nasal provocation test with D. farinae and/or D. pteronyssinus in allergic rhinitis patients sensitized to house dust mite
Cytokines in nasal lavage fluid | Baseline and 4 months after the first injection
  Cytokines of Th1, Th2, and Treg in nasal lavage fluid
Exhaled NO | Baseline and 4 months after the first injection
  Exhaled nitric oxide measuring NIOX MINO, Thermofisher Scientific, Sweden
Respiratory and dermatologic symptoms provoked by allergen exposure in daily life | Baseline and 4 months after the first injection
  Visual analogue scale of respiratory and dermatologic symptoms provoked by allergen exposure in daily life (ranged from 0 to 100)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Min Lee, M.D., Ph.D., Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Background] Zaleska A, Eiwegger T, Soyer O, van de Veen W, Rhyner C, Soyka MB, Bekpen C, Demiroz D, Treis A, Sollner S, Palomares O, Kwok WW, Rose H, Senti G, Kundig TM, Ozoren N, Jutel M, Akdis CA, Crameri R, Akdis M. Immune regulation by intralymphatic immunotherapy with modular allergen translocation MAT vaccine. Allergy. 2014 Sep;69(9):1162-70. doi: 10.1111/all.12461. Epub 2014 Jul 12. PMID 24934402
- [Result] Kundig TM, Johansen P, Bachmann MF, Cardell LO, Senti G. Intralymphatic immunotherapy: time interval between injections is essential. J Allergy Clin Immunol. 2014 Mar;133(3):930-1. doi: 10.1016/j.jaci.2013.11.036. Epub 2014 Jan 15. No abstract available. PMID 24439076
- [Result] Witten M, Malling HJ, Blom L, Poulsen BC, Poulsen LK. Is intralymphatic immunotherapy ready for clinical use in patients with grass pollen allergy? J Allergy Clin Immunol. 2013 Nov;132(5):1248-1252.e5. doi: 10.1016/j.jaci.2013.07.033. Epub 2013 Sep 13. No abstract available. PMID 24035151
- [Result] Senti G, Crameri R, Kuster D, Johansen P, Martinez-Gomez JM, Graf N, Steiner M, Hothorn LA, Gronlund H, Tivig C, Zaleska A, Soyer O, van Hage M, Akdis CA, Akdis M, Rose H, Kundig TM. Intralymphatic immunotherapy for cat allergy induces tolerance after only 3 injections. J Allergy Clin Immunol. 2012 May;129(5):1290-6. doi: 10.1016/j.jaci.2012.02.026. Epub 2012 Mar 30. PMID 22464647
- [Result] Senti G, Johansen P, Kundig TM. Intralymphatic immunotherapy: from the rationale to human applications. Curr Top Microbiol Immunol. 2011;352:71-84. doi: 10.1007/82_2011_133. PMID 21725898
- [Result] Senti G, Johansen P, Kundig TM. Intralymphatic immunotherapy. Curr Opin Allergy Clin Immunol. 2009 Dec;9(6):537-43. doi: 10.1097/ACI.0b013e3283310ff7. PMID 19680119
- [Result] Senti G, Prinz Vavricka BM, Erdmann I, Diaz MI, Markus R, McCormack SJ, Simard JJ, Wuthrich B, Crameri R, Graf N, Johansen P, Kundig TM. Intralymphatic allergen administration renders specific immunotherapy faster and safer: a randomized controlled trial. Proc Natl Acad Sci U S A. 2008 Nov 18;105(46):17908-12. doi: 10.1073/pnas.0803725105. Epub 2008 Nov 10. PMID 19001265
- [Result] Hylander T, Latif L, Petersson-Westin U, Cardell LO. Intralymphatic allergen-specific immunotherapy: an effective and safe alternative treatment route for pollen-induced allergic rhinitis. J Allergy Clin Immunol. 2013 Feb;131(2):412-20. doi: 10.1016/j.jaci.2012.10.056. PMID 23374268